CLINICAL TRIAL: NCT04596930
Title: MR-guided LITT Therapy in Patients With Primary Irresectable Glioblastoma: a Randomized Pilot Study
Brief Title: MR-guided LITT Therapy in Patients With Primary Irresectable Glioblastoma
Acronym: EMITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL73896.091.20
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LITT arm (Experimental): Patients will be randomized to receive biopsy and LITT (n=10)
  Interventions: Procedure: Laser ablation thermal therapy

INTERVENTIONS:
Procedure: Laser ablation thermal therapy — The Visualase Thermal Therapy System is used to necrotize or coagulate soft tissue through interstitial irradiation under MRI guidance

SUMMARY:
Objective: In preparation of a randomized controlled trial, the investigators aim to assess pilot data on technical feasibility and safety of laser interstitial thermal therapy (LITT) at Radboud University Medical centre and to assess practical feasibility of a randomized study in patients with primary irresectable glioblastoma, as compared with standard of care.

Study design: Prospective randomized pilot study. Randomization stopped (amendment September 2nd, 2021),

Study population: 20 patients aged >= 18 with radiologically suspected diagnosis of primary glioblastoma and contra-indication for surgical resection.

Intervention: Patients will be randomized to receive either (i) biopsy and LITT (n=10) or (ii) biopsy alone (n=10).

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in the study, a patient must meet all of the following criteria:

* Informed consent, age >18-year-old
* Supratentorial localization
* Maximal volume <=70cc on post-contrast T1 MRI
* Safe trajectory/trajectories possible for ablation of 70% of the tumour, avoiding eloquent structures or transgression of a ventricle or vessel .
* Karnofsky Performance Status (KPS) >= 70

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Contra-indication for general anaesthesia or MRI
* Lesion >70cc on post-contrast MRI on the day before intervention.
* Non-glioblastoma diagnosis as per frozen section analysis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Inclusion rate of patients meeting the inclusion criteria | 12 months
  To assess practical feasibility of a randomized study in this patient population, in preparation of a future randomized controlled trial
Number drop out (informed consent) | 30 days
  To assess practical feasibility of a randomized study in this patient population, in preparation of a future randomized controlled trial
Number of patients with completed follow-up at 3 months | 3 months
  To assess practical feasibility of a randomized study in this patient population, in preparation of a future randomized controlled trial
30-days mortality | 30 days
  To assess safety of LITT at our center in patients with irresectable glioblastoma
Number of patients with complications | 3 months
  To assess safety of LITT at our center in patients with irresectable glioblastoma
Time from inclusion to procedure | 3 months
  To assess feasibility of LITT at our center in patients with irresectable glioblastoma
Time from LITT to adjuvant therapy | 3 months
  To assess feasibility of LITT at our center in patients with irresectable glioblastoma
Ablation of 90 percent of the target lesion in at least 70 percent of patients | 3 months
  To assess feasibility of LITT at our center in patients with irresectable glioblastoma

SECONDARY OUTCOMES:
Overall survival and progression free survival | 12 months
  To assess preliminary data on survival
Euro quality of life-5D (from 11111, best outcome to 55555 worse outcome) | 3 months
  To assess preliminary data on quality of life
European Organisation for Research and Treatment of Cancer - BN20 brain module | 3 months
  To assess preliminary data on quality of life
Tumor volume evolution | 3 months
  To assess tumour volume evolution on MRI at 3 months post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud UMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viozzi I, Overduin CG, Rijpma A, Rovers MM, Laan MT. MR-guided LITT therapy in patients with primary irresectable glioblastoma: a prospective, controlled pilot study. J Neurooncol. 2023 Sep;164(2):405-412. doi: 10.1007/s11060-023-04371-x. Epub 2023 Jul 28. PMID 37505379